CLINICAL TRIAL: NCT01859741
Title: A Phase 1b/2 Study of OMP-59R5 in Combination With Etoposide and Platinum Therapy in Subjects With Untreated Extensive Stage Small Cell Lung Cancer (PINNACLE)
Brief Title: A Phase 1b/2 Study of OMP-59R5 (Tarextumab) in Combination With Etoposide and Platinum Therapy
Acronym: PINNACLE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: OMP-59R5 did not improve PFS.
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 59R5-003
Record Dates: First submitted 2013-05-16; First posted 2013-05-22 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Stage IV Small Cell Lung Cancer
Keywords: Newly diagnosed Stage IV Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — tarextumab; Etoposide; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OMP-59R5 Combination with Etoposide and Cisplatin (Experimental)
  Interventions: Drug: OMP-59R5; Drug: Etoposide; Drug: Placebo; Drug: Cisplatin or Carboplatin
- Etoposide and Cisplatin plus Placebo (Experimental)
  Interventions: Drug: OMP-59R5; Drug: Etoposide; Drug: Placebo; Drug: Cisplatin or Carboplatin

INTERVENTIONS:
Drug: OMP-59R5 — OMP-59R5 administered intravenously
  Other Names: Tarextumab
Drug: Etoposide — administered intravenously
Drug: Placebo — administered IV
Drug: Cisplatin or Carboplatin — administered intravenously

SUMMARY:
The study consists of a Phase1b lead-in portion to determine the maximum tolerated dose (MTD) of OMP-59R5 (tarextumab) in combination with etoposide (EP) for 6 cycles followed a Phase 2, multi center, randomized, placebo-controlled portion comparing the efficacy and safety of OMP-59R5 in combination with EP for 6 cycles followed by single agent OMP-59R5 relative to EP alone for 6 cycles in subjects receiving first-line therapy for extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
The Phase 1b lead-in portion of the study was conducted to determine the MTD of OMP-59R5 administered along with EP. The Phase 2 portion of the study was multi-center, randomized, and placebo-controlled. Subjects who qualified for enrollment into the Phase 2 portion of the study were randomized in a 1:1 ratio to receive study treatment of tarextumab along with EP (Arm A) or placebo along with EP (Arm B).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for the study:

1. Histologically or cytologically documented extensive stage small cell lung cancer.
2. Adults of 18 years of age or older.
3. Performance Status (ECOG) of 0 or 1.
4. Formalin Fixed Paraffin Embedded (FFPE) tumor tissue.
5. Adequate organ function:

   1. Adequate hematologic function (absolute neutrophil count [ANC] ≥ 1,500 cells/μL; hemoglobin ≥ 9 g/dL, platelets ≥ 100,000/μL).
   2. Adequate renal function (serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance ≥ 60 mL/min using Cockcroft-Gault formula).
   3. Adequate hepatic function (alanine aminotransferase [ALT] ≤ 3 x upper limit of normal [ULN], ALT may be ≤ 5 x ULN if due to liver metastases but cannot be associated with concurrent elevated bilirubin >1.5 times the upper limit of normal (ULN) unless it is approved by the Sponsor's Medical Monitor).
   4. Prothrombin Time (PT)/International Normalized Ration (INR) ≤1.5 × ULN, activated partial thromboplastin time (aPTT) ≤1.5 × ULN.
6. Written consent on an Institutional Review Board (IRB)/IndependentEthics Committee (IEC)-approved Informed Consent Form prior to any study-specific evaluation.
7. For women of child-bearing potential, negative serum pregnancy test at screening and use of physician-approved method of birth control from 30 days prior to the first study drug administration to 30 days following the last study drug administration or the last EP in the study, whichever is discontinued last.
8. Male subjects must be surgically sterile or must agree to use physician-approved contraception during the study and for 30 days following the last study drug administration or the last EP in the study, whichever is discontinued last.

Exclusion Criteria:

Subjects who meet any of the following criteria will not be eligible for participation in the study:

1. Limited stage small cell lung cancer appropriate for radical treatment with chemoradiation.
2. Prior therapy including radiation, chemotherapy or surgery for newly diagnosed extensive stage small cell lung cancer.
3. Presence of any serious or uncontrolled illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure unstable angina pectoris, uncontrolled cardiac arrhythmia, uncontrolled arterial thrombosis, symptomatic pulmonary embolism, and psychiatric illness that would limit compliance with study requirement.
4. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty and/or stenting within 6 months prior to the first administration of study drug.
5. A history of malignancy with the exception of:

   1. Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer
   2. Adequately treated stage I cancer from which the subject is currently in remission, or
   3. Any other cancer from which the subject has been disease-free for ≥ 3 years
6. Known human immunodeficiency virus (HIV) infection.
7. Females who are pregnant or breastfeeding.
8. Concurrent use of therapeutic warfarin (prophylactic low dose of warfarin, i.e., 1 mg daily for port catheter is allowed)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2012-01-07 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Highlands Oncology Group, Rogers, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Sarah Cannon, Fort Myers, Florida
  - Ocala Oncology Center, PL, Ocala, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Georgia Cancer Specialists, PC, Atlanta, Georgia
  - Univeristy of Chicago Medical Center, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Weinberg Cancer Institute, Baltimore, Maryland
  - University of Michigan Medical Center, Clinical Trials Office, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology Hematology , P.A., Minneapolis, Minnesota
  - Oncology Hematology West PC, dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Providence Cancer Center Oncology and Hematology Care Eastside, Portland, Oregon
  - UPMC Cancer Pavilion, Pittsburgh, Pennsylvania
  - Greenville Health System, Clinical Research Unit, Institute for Translational Oncology Research, Greenville, South Carolina
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology-South Austin, Austin, Texas
  - Texas Oncology-Bedford, Bedford, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - The University of Texas MD A nderson Cancer Center, Houston, Texas
  - Cancer Care Network of South Texas, San Antonio, Texas
  - Oncology and Hematology Associates of Southwest Virginia Inc., Blacksburg, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1b: Approximately 30 subjects were planned. A total of 27 subjects were enrolled.
  Phase 2: Approximately 135 subjects were planned to be randomized. A total of 145 subjects were enrolled/randomized.
  Total: 172 subjects were enrolled/randomized (Phase 1b and Phase 2)
Groups:
- P1B: OMP-59R5 5mg/kg + ETO + CIS: Cohort 1: Subjects receive OMP-59R5 5 mg/kg (administered on Day 1 of each 21-day cycle) along with etoposide 100 mg/m2 (Days 1, 2, and 3) and cisplatin 80 mg/m2 (Day 1).
- P1B: OMP-59R5 7.5 mg/kg + ETO + CIS: Cohort 2: Subjects receive OMP-59R5 7.5 mg/kg (administered on Day 1 of each 21-day cycle) along with etoposide 100 mg/m2 (Days 1, 2, and 3) and cisplatin 80 mg/m2 (Day 1).
- P1B: OMP-59R5 10 mg/kg + ETO + CIS: Cohort 3: Subjects receive OMP-59R5 10 mg/kg (administered on Day 1 of each 21-day cycle) along with etoposide 100 mg/m2 (Days 1, 2, and 3 and cisplatin 80 mg/m2 on Day 1).
- P1B: OMP-59R5 12.5 mg/kg + ETO + CIS: Cohort 4: Subjects receive OMP-59R5 12.5 mg/kg (administered on Day 1 of each 21-day cycle) along with etoposide 100 mg/m2 (Days 1, 2, and 3) and cisplatin 80 mg/m2 (Day 1).
- P1B: OMP-59R5 15 mg/kg + ETO + CIS: Cohort 5: Subjects receive OMP-59R5 15 mg/kg (administered on Day 1 of each 21-day cycle) along with etoposide 100 mg/m2 (Days 1, 2, and 3) and cisplatin 80 mg/m2 (Day 1).
- P1B: OMP-59R5 15mg/kg + ETO + CARB: Cohort 6: Subjects receive OMP-59R5 15 mg/kg (administered on Day 1 of each 21-day cycle) along with etoposide 100 mg/m2 (Days 1, 2, and 3) and carboplatin AUC of 5 mg/mL•min (Day 1).
- P2: Placebo + CIS or CARB: Placebo Arm: Active Arm: Subjects receive placebo and etoposide 100 mg/m2 and cisplatin 75 mg/m2 or carboplatin AUC 5 mg/kg *min
- P2: OMP-59R5 15 mg/kg + ETO and CIS or CARB: Active Arm: Subjects receive OMP-59R5 15 mg/kg and etoposide 100 mg/m2 and cisplatin 75 mg/m2 or carboplatin AUC 5 mg/kg *min
Period: Overall Study
Arm/Group | P1B: OMP-59R5 5mg/kg + ETO + CIS | P1B: OMP-59R5 7.5 mg/kg + ETO + CIS | P1B: OMP-59R5 10 mg/kg + ETO + CIS | P1B: OMP-59R5 12.5 mg/kg + ETO + CIS | P1B: OMP-59R5 15 mg/kg + ETO + CIS | P1B: OMP-59R5 15mg/kg + ETO + CARB | P2: Placebo + CIS or CARB | P2: OMP-59R5 15 mg/kg + ETO and CIS or CARB
Started | 3 | 3 | 6 | 3 | 6 | 6 | 72 | 73
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Not Completed | 3 | 3 | 6 | 3 | 6 | 6 | 70 | 70
Not completed — Death | 3 | 2 | 4 | 3 | 5 | 4 | 51 | 51
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 1 | 0 | 16 | 14
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | P1B: OMP-59R5 5mg/kg + ETO + CIS | P1B: OMP-59R5 7.5 mg/kg + ETO + CIS | P1B: OMP-59R5 10 mg/kg + ETO + CIS | P1B: OMP-59R5 12.5 mg/kg + ETO + CIS | P1B: OMP-59R5 15 mg/kg + ETO + CIS | P1B: OMP-59R5 15mg/kg + ETO + CARB | P2: OMP-59R5 15 mg/kg + ETO and CIS or CARB | P2: Placebo + CIS or CARB | Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 6 | 6 | 73 | 72 | 172
Age, Customized [Mean (Full Range); unit: years]
  Age | 68.3 [59 to 83] | 72.3 [65 to 84] | 67.7 [59 to 72] | 64.3 [51 to 73] | 61.0 [53 to 67] | 57.2 [40 to 78] | 65.3 [40 to 81] | 65.4 [33 to 83] | 58.5 [33 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 0 | 3 | 3 | 30 | 37 | 77
  Male | 2 | 2 | 4 | 3 | 3 | 3 | 43 | 35 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 6 | 13
  White | 3 | 3 | 6 | 3 | 6 | 4 | 66 | 64 | 155
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 3 | 6 | 6 | 73 | 72 | 172

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: To Determine the Maximum Tolerated Dose (MTD) of OMP-59R5 When Administered With Etoposide and Cisplatin or Carboplatin (Number of Subjects With DLTs)
Description: To determine the MTD of tarextumab when administered on Day 1 of each 21 day cycle along with etoposide 100 mg/m2 on Days 1, 2 and 3, and cisplatin 80 mg/m2 or carboplatin area under the curve (AUC) of 5 mg/mL•min on Day 1 in subjects with untreated extensive stage small cell lung cancer. DLT evaluable population includes all subjects who received at least 1 partial dose of OMP-59R5 during the Phase 1b dose escalation portion of the study including the carboplatin cohort and who had completed Day 21 cycle of 1 OMP-59R5 administration or had discontinued due to drug-related toxicity.
Time Frame: Up to 1 year in absence of unacceptable toxicity or disease progression.
Population: The MTD of OMP-59R5 in combination with etoposide and cisplatin or carboplatin was not reached and the recommended phase 2 dose was determined to be 15 mg/kg every 21-day cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | P1B: OMP-59R5 5mg/kg + ETO + CIS | P1B: OMP-59R5 7.5 mg/kg + ETO + CIS | P1B: OMP-59R5 10 mg/kg + ETO + CIS | P1B: OMP-59R5 12.5 mg/kg + ETO + CIS | P1B: OMP-59R5 15 mg/kg + ETO + CIS | P1B: OMP-59R5 15mg/kg + ETO + CARB
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 6 | 6
Participants | 0 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Phase 1b: Overall Response (Response Evaluable Population)
Description: The best overall response is defined as the best Investigator-assessed response recorded from the start of the treatment until disease progression in the following order of importance: Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), Not Evaluable (NE). Response evaluable population includes subjects who received 1 partial dose of OMP-59R5 and at at least 1 post tumor assessment.
Time Frame: Up to 1 year in absence of unacceptable toxicity or disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | P1B: OMP-59R5 5mg/kg + ETO + CIS | P1B: OMP-59R5 7.5 mg/kg + ETO + CIS | P1B: OMP-59R5 10 mg/kg + ETO + CIS | P1B: OMP-59R5 12.5 mg/kg + ETO + CIS | P1B: OMP-59R5 15 mg/kg + ETO + CIS | P1B: OMP-59R5 15mg/kg + ETO + CARB
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 6 | 6
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 3 | 2 | 4 | 2 | 5 | 4
  Stable Disease | 0 | 1 | 1 | 1 | 0 | 1
  Progressive Disease | 0 | 0 | 0 | 0 | 1 | 1
  Not Evaluated | 0 | 0 | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Phase 2: Progression Free Survival (ITT Population)
Description: To determine the improvement in Progression Free Survival (PFS) resulting from the addition of tarextumab to etoposide and platinum therapy (EP) in subjects receiving first-line therapy for extensive stage small cell lung cancer. PFS is based on the Investigator-assessments of tumor response which is defined as the number of days from randomization until death or disease progression as defined by RECIST criteria for the ITT Population.
Time Frame: Up to 1 year until disease progression or death.
Measure: Count of Participants; unit: Participants
Arm/Group | P2: Placebo + CIS or CARB | P2: OMP-59R5 15 mg/kg + ETO and CIS or CARB
Number analyzed (Participants) | 72 | 73
Participants
  Disease Progression or Death | 56 | 51
  Did not Progress or Die | 16 | 22

4. Primary Outcome: Phase 2: Best Overall Tumor Response Based on Investigator Assessment (ITT Population)
Description: The response rate is the number of subjects per treatment arm who have either a complete response (CR) or partial response (PR) for best overall response (according to RECIST criteria) divided by the number of subjects randomized to the respective arms.
Time Frame: Up to 1 year in absence of unacceptable toxicity or disease progression
Measure: Count of Participants; unit: Participants
Arm/Group | P2: Placebo + CIS or CARB | P2: OMP-59R5 15 mg/kg + ETO and CIS or CARB
Number analyzed (Participants) | 72 | 73
Participants
  Complete Response | 2 | 1
  Partial Response | 49 | 49
  Stable Disease | 10 | 9
  Progressive Disease | 4 | 2
  Not Evaluable | 1 | 1
  No Post-Baseline Tumor Assessment Collected | 6 | 11

ADVERSE EVENTS:
Time Frame: Adverse event and serious adverse event data are collected from the time of first administration of OMP-59R5, etoposide or platinum therapy up to 4 weeks after the last administration OMP-59R5, etoposide or platinum therapy, whichever is discontinued last but but before the initiation of a new anti-cancer therapy. All cause mortality was collected every 3 months until death, loss to follow-up or study termination by the sponsor (up to 35 months).
Description: P1: All cause mortality was assessed on the ITT population which was comprised of all subjects who receive at least one partial dose of OMP-59R5. Serious and non-serious AEs were assessed on the ITT population.
  P2: All cause mortality was assessed on the ITT population which was comprised of all randomized subjects. Serious and non-serious AEs were assessed on the Safety Population which was defined as all subjects who received one partial dose of OMP-59R5 or placebo.
Arm/Group | P1B: OMP-59R5 5mg/kg + ETO + CIS | P1B: OMP-59R5 7.5 mg/kg + ETO + CIS | P1B: OMP-59R5 10 mg/kg + ETO + CIS | P1B: OMP-59R5 12.5 mg/kg + ETO + CIS | P1B: OMP-59R5 15 mg/kg + ETO + CIS | P1B: OMP-59R5 15mg/kg + ETO + CARB | P2: Placebo + CIS or CARB | P2: OMP-59R5 15 mg/kg + ETO and CIS or CARB
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3 | 4/6 | 3/3 | 5/6 | 4/6 | 51/72 | 51/73
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 6/6 | 1/3 | 0/6 | 3/6 | 29/68 | 37/69
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 3/3 | 6/6 | 6/6 | 68/68 | 69/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P1B: OMP-59R5 5mg/kg + ETO + CIS (N=3) | P1B: OMP-59R5 7.5 mg/kg + ETO + CIS (N=3) | P1B: OMP-59R5 10 mg/kg + ETO + CIS (N=6) | P1B: OMP-59R5 12.5 mg/kg + ETO + CIS (N=3) | P1B: OMP-59R5 15 mg/kg + ETO + CIS (N=6) | P1B: OMP-59R5 15mg/kg + ETO + CARB (N=6) | P2: Placebo + CIS or CARB (N=68) | P2: OMP-59R5 15 mg/kg + ETO and CIS or CARB (N=69)
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 12
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | P1B: OMP-59R5 5mg/kg + ETO + CIS (N=3) | P1B: OMP-59R5 7.5 mg/kg + ETO + CIS (N=3) | P1B: OMP-59R5 10 mg/kg + ETO + CIS (N=6) | P1B: OMP-59R5 12.5 mg/kg + ETO + CIS (N=3) | P1B: OMP-59R5 15 mg/kg + ETO + CIS (N=6) | P1B: OMP-59R5 15mg/kg + ETO + CARB (N=6) | P2: Placebo + CIS or CARB (N=68) | P2: OMP-59R5 15 mg/kg + ETO and CIS or CARB (N=69)
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 5 | 3 | 5 | 6 | 23 | 53
Nausea (Gastrointestinal disorders) | 3 | 2 | 4 | 2 | 4 | 4 | 44 | 36
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4 | 1 | 3 | 3 | 11 | 22
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 2 | 1 | 28 | 11
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 8 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 6 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 4
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Perianal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 3 | 2 | 3 | 2 | 16 | 26
Hypercreatininaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 4 | 1 | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 3 | 1 | 15 | 15
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 3 | 1 | 1 | 2 | 14 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 5 | 24
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 4 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 9 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 9
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 2 | 1 | 3 | 4 | 38 | 35
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 4 | 1 | 4 | 3 | 12 | 40
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1 | 3 | 0 | 32 | 22
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 5
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 10 | 6
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4
Fatigue (General disorders) | 3 | 3 | 3 | 2 | 5 | 1 | 43 | 43
Oedema peripheral (General disorders) | 3 | 1 | 1 | 1 | 2 | 2 | 13 | 8
Pyrexia (General disorders) | 2 | 0 | 0 | 1 | 1 | 1 | 8 | 5
Asthenia (General disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 7 | 10
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 9
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 6
Device occlusion (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 3 | 1 | 7 | 8
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 2 | 1 | 13 | 14
Dysgeusia (Nervous system disorders) | 0 | 0 | 3 | 1 | 0 | 1 | 7 | 13
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 5 | 3
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 4
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 2 | 2 | 18 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 17 | 14
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 5 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 5 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 2 | 4 | 2 | 27 | 27
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 2 | 1 | 3 | 0 | 1 | 1 | 11 | 18
Basophil count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 9
Blood bilirubin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 2 | 4 | 13
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 4
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Corneal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 11 | 8
Vulval abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 10 | 9
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 10 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 7 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 3 | 0 | 1 | 1 | 7 | 5
Depression (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 7
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 8 | 13
Hypotension (Vascular disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 10 | 5
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 6 | 6
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 5 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 3
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 1 | 3 | 3
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 11
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
Infusion site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 7
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urea decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram ST segment abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine ketone body present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood sodium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypohidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conduction disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blindness unilateral (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT01859741/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT01859741/Prot_ICF_001.pdf